CLINICAL TRIAL: NCT02605239
Title: Effect on Oral Health, Phycosocial Impact and Esthetics Perception of Bleaching Teeth
Brief Title: Phycosocial Impact of Bleaching Teeth
Acronym: PSYBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof. Dr. Eduardo Fernández, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-18a
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration | interventions — Tooth Bleaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bleaching teeth (Experimental): Group of patients will be bleaching with 10% peroxide carbamide , and them will be assessed the impact on dental confidence , impact psychosocial and esthetic perception
  Interventions: Drug: Bleaching teeth

INTERVENTIONS:
Drug: Bleaching teeth — bleaching teeth with carbamide peroxide 10% for 3 weeks
  Other Names: bleaching gel

SUMMARY:
58 patients between 18 and 76 years who attended the Operative Dentistry Clinic at Dental School, Universidad de Chile, were included in the study. Those patients were bleaching and included in this study and signed a consent form. The patients were treated with 10% carbamide peroxide (CP) gel (Whiteness Perfect, FGM) to each subject with verbal instructions for 3 weeks with daily applications of 1 hour according to manufacturers indications , before and after this procedure was applied again the OHIP-Esthetics , PIDAQ and OES questionnaire form, had 30 minutes to answer it, were completed before , immediately after and one month control post-bleaching procedure.

DETAILED DESCRIPTION:
This study was approved by the Ethics Committee of the Faculty of Dentistry (13/18a). This study included 58 patients aged between 18 and 76 years who attended the Operative Dentistry Clinic at the Dental School from the Local University and were eligible for bleaching (see eligibility criteria in the next item). Dental bleaching, free of charge, was suggested to the patients as a way to improve the patient's smile. The patients were informed about the benefits and possible side effects of the procedure in a standardized manner.

Eligibility criteria for dental bleaching Participants were evaluated in a dental chair and after prophylactic dental treatment with pumice and water. To be eligible for dental bleaching, participants should have good general and oral health. Each subject should have at least one central incisor shaded A2 or darker, assessed by comparison with a value-oriented shade guide (Vita classical; Vita Zahnfabrik, Bad Säckingen, Germany). Patients who had undergone previous dental bleaching procedures, under orthodontic treatment, who were pregnant or lactating, or who had bruxism habits were not eligible for dental bleaching. Participants with restorations on the labial surfaces of their anterior teeth, non-carious cervical lesions, veneers, full crowns, gingival recession, spontaneous tooth pain, internal tooth discoloration, and teeth with endodontic treatment or fluorosis were also not included as they could not be immediately eligible for dental bleaching.

Bleaching Procedure For the participants who were bleaching procedure, we made alginate impressions of each subject's maxillary and mandibular arches, and these were filled with dental stone. We did not apply block-out material to the labial surfaces. A 1-mm soft vinyl material, provided by the manufacturer (FGM Dental Products, Joinville, SC, Brazil) was used to fabricate the custom-fitted tray to hold the bleaching gel. The bleaching tray was trimmed 1 mm beyond the marginal gingiva and we delivered a 10% carbamide peroxide (CP) gel (Whiteness Perfect, FGM) to each participant. We give them verbal instructions to apply the product 1 hour daily for 3 weeks. After each application, the patient should remove the tray, wash it with water, and brush teeth as usual. Verbal instructions for oral hygiene were also given, encouraging regular brushing with fluoridated toothpastes that did not contain whitening components.

For these participants, the OHIP-Esthetics, PIDAQ and OES surveys were applied before , one week and one month after the end of the bleaching procedure, and the patient was also given 30 minutes to complete it.

Color Evaluation Color evaluations were performed using subjective and objective methods. For the subjective evaluation, the 16 tabs of the Vita shade Classical guide Vita classical (Vita Zahnfabrik, Bad Säckingen, Germany) were arranged from highest (B1) to lowest (C4) value and used to determine tooth color. Although this scale is not linear in the truest sense, it was treated as continuous with a linear ranking. Two calibrated evaluators with an agreement of at least 85% (using weighted kappa statistics) recorded the shade of the middle area of the labial surface of the upper central right incisor according to the American Dental Association guidelines. Color was registered at baseline and during treatment (after the first, second, and third week of bleaching), and one week and one month after the end of the bleaching protocol to corroborate the effectiveness of bleaching procedure. The color change between baseline and each recall time was calculated as the change in the number of shade guide units (ΔSGU), which occurred toward the lightest end of the value-oriented list of shade tabs. In case the operators disagreed on the color, a consensus was reached before dismissing the patient.

In the objective evaluation, a digital spectrophotometer (Vita Easyshade, Vita Zahnfabrik) with a reliability of 97% was used. An impression of the maxillary arch was taken with dense silicone paste (Coltoflax and Perfil Cub, Vigodent, Rio de Janeiro, Brazil) and a window was created on the labial surface of the silicone guide using a metal device with a radius of 6 mm to allow adaptation of the tip of the spectrophotometer device and to standardize the spectrophotometric color evaluation across all recall periods.

The color coordinates (L*, a*, and b*) were recorded. The value for L* represented the value from 0 (black) to 100 (white), and a* and b* represented color along the red-green axis and yellow-blue axis, respectively. The difference between baseline and each recall period (∆E) was calculated using the formula (CIE, 1978) ∆E = [(∆L*)2+(∆a*)2+(∆b*)2]1/2.

Tooth Sensitivity Evaluation Patients were asked to keep a daily record of whether they experienced tooth sensitivity (TS). The participants were instructed to indicate their daily pain using a visual analog scale (VAS).3, 6, 7 This scale is a 10-cm horizontal line labeled no tooth sensitivity at one end and unbearable tooth sensitivity at the other end. The patient should mark with a vertical line across the horizontal line of the scale the intensity of the tooth sensitivity. Then, the distance in mm from the zero end was measured with the aid of a millimeter ruler.

Oral Health Impact Profile (OHIP-Esthetics) questionnaire Satisfaction was measured using the OHIP-Esthetics questionnaire validated in Chilean Spanish .The questionnaire was administered by a research operator at baseline, at one week, one month and nine months (before prophylaxis) after bleaching. Each statement was accompanied by a Likert-type scale, which generated a score ranging from 4 to 0 (very often = 4, fairly often = 3, occasionally = 2, hardly never = 1, never = 0). These individual scores were added together to give a summary score ranging from 0 (minimum) to 56 (maximum). The outcomes were considered the sum of the OHIP-Esthetics and dimension scores. The internal consistency was evaluated using Cronbach's Alpha test.

The Psychosocial Impact of Dental Esthetics Questionnaire (PIDAQ) questionnaire The questionnaire consisted of 23 items grouped into four components using factor analysis: 1) dental self-confidence ; 2) social impact ; 3) psychosocial impact ; and 4) esthetic concern .9 The first factor, dental self-confidence, consisted of six items from the self-confidence scale. The second factor, social impact, contained eight items from the social aspects scale of the quality of life questionnaire. The third factor, psychosocial impact, was derived from six formulated items relating mainly to the psychosocial impact of dental esthetics. The fourth factor was the esthetics. The patient was asked to evaluate the items using a five-point Likert scale with numerical values 0 = "not at all", 1 = "a little", 2 = "somewhat", 3 = "strongly" and 4 = "very strongly". The questionnaire was administered by a research operator at baseline, one week, one month, and nine months (before prophylaxis) after bleaching and was validated in Spanish with a confidence reported by Cronbach´s alpha of 0.90.10 The outcomes were considered the sum of the PIDAQ questionnaire and factor scores; the internal consistency was evaluated using the Cronbach's Alpha test.

Orofacial Esthetic Scale (OES) The Orofacial Esthetic Scale was originally developed in the Swedish language, the OES-S. For international use, the OES-S was translated into English,resulting in the OES-E . The OES consists of eight questions, assessing the appearance of the face, profile, mouth, tooth alignment, tooth shape, tooth colour and gums, as well as an overall impression of oro-facial aesthetics. Answers to the eight questions are scored on 11-point numeric rating scales, ranging from 'Very dissatisfied' (score 0) to 'Very satisfied' (score 10). The scores of the first seven items are added to a summary score. Therefore, the OES summary score ranges from 0 (worst score -patient is very dissatisfied with all aesthetics items) up to 70 (best score - patient is very satisfied with all aesthetics items). The score of the eighth item (overall impression score) is judged separately, thus ranging from 0 (worst score - patient is very dissatisfied on global assessment) up to 10 (best score - patient is very satisfied on global assessment). Hence, lower scores imply more impaired self-perceived oro-facial aesthetics.

Sample size calculation Based on previous study we considered a difference of 4 units in any of the domains to be clinically important. With a significance level of 5% and a power of 90%, a minimum sample size of 58 participants per group would be required to detect a difference of 4 units in one of the domains of the questionnaires on before and after comparisons.

Data collection and statistical analysis Data from the OHIP-Esthetics PIDAQ and OES were collected on a spreadsheet and analyzed by a psychologist that was blind to the group assignment.

Normality of the data bleaching and the homogeneity of the variance-covariance matrix were evaluated with the Kolmogórov-Smirnov test. As data was not normally distributed, treatment efficacy (ΔE and ΔSGU) was evaluated with respect to color change using the Wilcoxon Signed Rank test.

The mean intensity of tooth sensitivity in VAS scale was reported as mean and standard deviations. The percentage of patients who experienced tooth sensitivity at least once during the bleaching therapy was considered the absolute risk of tooth sensitivity, reported as percentage with the 95% confidence interval.

All statistical analyses were performed using SPSS 22.0 (SPSS Inc., Chicago, IL, USA) at a level of significance of 5% (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with Anterior teeth without restorations, previous bleaching procedures, cervical lesions, or dental pain

Exclusion Criteria:

* Pregnant or lactating,
* Had moderate or severe fluorosis,
* Tetracycline stains,
* Orthodontic treatment,
* Periodontal disease,
* Orofacial tumors,
* Trauma,
* Tooth malformation Were taking analgesic, anti-inflammatory, or antibiotic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Oral Health and quality of Life | 1 month
  Assesed by OHIP-Esthetics survey

SECONDARY OUTCOMES:
phycosocial impact | 1 month
  Assesed by PIDAQ survey
esthetics perception | 1 month
  Assesed by OES survey

CONTACTS AND LOCATIONS:
Overall Officials: eduardo fernandez, Study Director — University of Chile
Locations (1):
- Eduardo Fernandez Godoy, Santiago, Chile

REFERENCES:
- [Background] Martin J, Vildosola P, Bersezio C, Herrera A, Bortolatto J, Saad JR, Oliveira OB Jr, Fernandez E. Effectiveness of 6% hydrogen peroxide concentration for tooth bleaching-A double-blind, randomized clinical trial. J Dent. 2015 Aug;43(8):965-72. doi: 10.1016/j.jdent.2015.05.011. Epub 2015 Jun 6. PMID 26057085
- [Derived] Bersezio C, Martin J, Herrera A, Loguercio A, Fernandez E. The effects of at-home whitening on patients' oral health, psychology, and aesthetic perception. BMC Oral Health. 2018 Dec 11;18(1):208. doi: 10.1186/s12903-018-0668-2. PMID 30537968